CLINICAL TRIAL: NCT00506103
Title: The No-Tie Technique Using the Harmonic Scalpel in Total Thyroidectomy With Central Neck Dissection: A Prospective Randomized Study
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Other Study IDs: SCHHN
Record Dates: First submitted 2007-07-21; First posted 2007-07-25 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: Hemorrhage; Hypocalcemia; Vocal Cord Palsy
Keywords: Thyroidectomy; Central neck dissection; Harmonic scalpel; Perioperative complications
MeSH Terms: conditions — Hemorrhage; Hypocalcemia; Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the safety and efficacy of the no-tie technique using the harmonic scalpel (HS) in terms of the operating time and complications in total thyroidectomy with central neck dissection (CND). Recently, the HS has been used as an alternative to conventional hand-tied ligation for hemostasis in thyroid surgery, which is a time-consuming procedure. Very limited data have been published on evidence of its safety in total thyroidectomy accompanied by CND without supplementary hand-tied ligation.

ELIGIBILITY:
Inclusion Criteria:

* patients with total thyroidectomy plus central neck dissection
* if primary tumor size was more than 1 cm in papillary thyroid cancer
* there was any evidence of lymph node enlargement in paratracheal lymph node group preoperatively or intraoperatively
* patients who underwent minimal resection of the surrounding soft tissues, including the sternothyroid or sternohyoid muscle, for extracapsular extension of thyroid cancer

Exclusion Criteria:

* patients who required lateral compartment neck dissection or mediastinal dissection for preexisting lymph node metastasis
* patients had clinical or laboratory indicators of coagulation disorders
* patients with preexisiting vocal cord palsy, fixation of the tumor to the recurrent laryngeal nerve requiring trnasection of the nerve
* patients with massive extracapsular extension to the surrounding soft tissues.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Woo Koh, MD, Principal Investigator — Dept. of Otolaryngology-Head and Neck Surgery, Soonchunhyang University College of Medicine
Locations (1):
- Dept. of otolaryngology-Head and Neck Surgery, Soonchunhyang University College of Medicine, Bucheon-si, South Korea

REFERENCES:
- [Background] Cordon C, Fajardo R, Ramirez J, Herrera MF. A randomized, prospective, parallel group study comparing the Harmonic Scalpel to electrocautery in thyroidectomy. Surgery. 2005 Mar;137(3):337-41. doi: 10.1016/j.surg.2004.09.011. PMID 15746789